CLINICAL TRIAL: NCT04984317
Title: Feasibility of Onabotulinumtoxin A Injection on Improving Female Stress Urinary Incontinence
Brief Title: Feasibility of BOTOX Injection on Improving Female Stress Urinary Incontinence
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Principal Investigator changing locations.
Sponsor: Northwell Health (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-04021756
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Botox Injection (Experimental): One-time injection of 100U BOTOX (onabotulinumtoxin A) into the fundus of the bladder under direct visualization via cystoscopy.
  Interventions: Drug: onabotulinumtoxin A

INTERVENTIONS:
Drug: onabotulinumtoxin A — One-time injection of 100U BOTOX
  Other Names: BOTOX

SUMMARY:
The purpose of this study is to assess the effect of onabotulinumtoxin A (BOTOX) injection into the detrusor muscle on increasing bladder compliance to reduce urinary leakage in women suffering from stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
The study involves a single-time injection of 100 units of onabotulinumtoxin A into the detrusor muscle of the bladder. Cystoscopy, which is the insertion of a scope with a small camera inside a tube into the participant's urethra. Then the doctor fills the participant's bladder with water or saline and sees detailed images of the injection site in the bladder while administrating the injection.

ELIGIBILITY:
Inclusion Criteria:

* Must be female sex and at least 18 years of age.
* Must be willing and able to complete all procedures and follow-up visits indicated in the protocol.
* Must have confirmed stress urinary incontinence (SUI) through urodynamic studies.
* Must have failed two non-invasive incontinence therapies (such as behavior modification, Kegel exercises, etc) for > 3 months.

Exclusion Criteria:

* Currently suffering from active urogenital infection.
* Has incontinence due to neurogenic causes (such as multiple sclerosis, cerebrovascular accident, spinal cord/brain injury, Parkinson Disease, detrusor-external sphincter dyssynergia, or similar conditions).
* Having concomitant pelvic floor or cystoscopic procedure.
* Has had prior surgical SUI treatment.
* Has had prior radiation therapy or brachy therapy.
* Has an atonic bladder or post-void residual (PVR) above 100cc on two or more occasions.
* Is pregnant or planning to become pregnant during the study duration.
* Has a contraindication to therapeutic BOTOX injections or cystoscopic procedures.
* Is enrolled in a concurrent clinical trial of any treatment (drug or device) that could affect urinary continence or bladder function without the sponsor's approval.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in the amount of urinary leakage post-treatment compared to baseline. | Baseline, 1-month, 3-month, 6-month
  1-hour pad weight, in grams

SECONDARY OUTCOMES:
Safety of 100U BOTOX injection as measured by the number of procedure-related adverse events. | Time of Procedure
  Adverse events may include organ perforation, bleeding, pelvic pain, infection, de novo dyspareunia, urinary retention, recurrent incontinence, other urinary problems and neuromuscular problems
Safety of 100U BOTOX injection as measured by the number of procedure-related adverse events. | 1-month
  Adverse events may include organ perforation, bleeding, pelvic pain, infection, de novo dyspareunia, urinary retention, recurrent incontinence, other urinary problems and neuromuscular problems
Safety of 100U BOTOX injection as measured by the number of procedure-related adverse events. | 3-month
  Adverse events may include organ perforation, bleeding, pelvic pain, infection, de novo dyspareunia, urinary retention, recurrent incontinence, other urinary problems and neuromuscular problems
Safety of 100U BOTOX injection as measured by the number of procedure-related adverse events. | 6-month
  Adverse events may include organ perforation, bleeding, pelvic pain, infection, de novo dyspareunia, urinary retention, recurrent incontinence, other urinary problems and neuromuscular problems
Change in patient-reported symptoms of stress incontinence symptoms via PGI-I. | 1-month, 3-month, 6-month
  The Patient Global Impression of Improvement (PGI-I) scale is a scale that measures improvement in symptoms and ranges from 1-7, with 1 indicating very much improvement and higher scores indicating less improvement.
Change in quality of life impacted by urinary incontinence via UDI-6. | Baseline, 1-month, 3-month, 6-month
  The Urinary Distress Inventory (UDI-6) is an inventory that assess symptoms and urinary incontinence and its severity on a scale of 0 to 3, with higher scores indicating greater symptom severity. IIQ-7 is a 30-item self-report questionnaire on the impact of urinary incontinence on activities roles and emotional states. Assigned values of the questionnaire are 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly.
Change in quality of life impacted by urinary incontinence via IIQ-7. | Baseline, 1-month, 3-month, 6-month
  The Incontinence Impact Questionnaire (IIQ-7) is a 30-item self-report questionnaire on the impact of urinary incontinence on activities roles and emotional states. Assigned values of the questionnaire are 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly.
Assessment of patient satisfaction post-treatment via SSQ-8. | 1-month
  The Surgical Satisfaction Questionnaire (SSQ-8) is a questionnaire about patient satisfaction after a surgery/procedure. Responses range from "Very unsatisfied" to "Very Satisfied".
Change in pain post-treatment compared to baseline via VAS. | Baseline, Time of Procedure, 1-month
  Scores are measured on a 100mm Visual Analog Scale (VAS). The VAS ranges from 0 to 100 with 0 indicating no pain and higher scores indicating greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No